CLINICAL TRIAL: NCT03587623
Title: Copeptin Serum Level in Liver Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Beata Błaszczyk, Principal Investigator, Medical University of Warsaw
Other Study IDs: Livercopeptin
Record Dates: First submitted 2018-07-03; First posted 2018-07-16 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Liver Cirrhosis; Copeptin; Liver Transplant
MeSH Terms: conditions — Liver Cirrhosis; Diabetes Insipidus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The study aim is to measure perioperative copeptin concentration in blood of liver transplant recipients and to assess whether there is a correlation between its level and hemodynamic derangement.

ELIGIBILITY:
Inclusion Criteria:

- Patient undergoing liver transplantation

Exclusion Criteria:

* Serum creatinine > 1,5 mg/dl
* Retransplantation
* Patient refusal
* CRRT or dialysis preoperatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing liver transplant
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2018-07-04 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Serum Copeptin concentration | Baseline, intraoperatively, 1,3,7,21 day postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- I Klinika Anestezjologii WUM, Warsaw, Mazovian Voivodeship, Poland